CLINICAL TRIAL: NCT05841394
Title: A Multi-center, Double-blinding, Parallel and Positive-controlled Phase III Clinical Trial for Efficacy and Safety Evaluation of Ilaprazole Sodium for Injection on Treatment of Prevention of Stress Ulcer Bleeding (Ilaprazole i.v. vs Esomeprazole, i.v.)
Brief Title: A Multi-center, Double-blinding, Parallel and Positive-controlled Phase III Clinical Trial for Efficacy and Safety Evaluation of Ilaprazole Sodium for Injection on Prevention of Stress Ulcer Bleeding
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Livzon Pharmaceutical Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LZ1075
Record Dates: First submitted 2023-04-22; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2022-08

CONDITIONS: Stress Ulcer Bleeding
MeSH Terms: interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esomeprazole Sodium (Active Comparator): 40 mg twice daily (q12h)
  Interventions: Drug: Esomeprazole 40mg; Drug: Placebo 2
- Ilaprazole Sodium (Experimental): 10 mg once daily, 20 mg dosed in the first day.
  Interventions: Drug: Ilaprazole Sodium; Drug: Placebo 1

INTERVENTIONS:
Drug: Esomeprazole 40mg — 40 mg i.v. twice daily (q12h)
  Arms: Esomeprazole Sodium
Drug: Ilaprazole Sodium — 10 mg i.v. once daily, 20 mg i.v. in the first day.
  Arms: Ilaprazole Sodium
Drug: Placebo 1 — Physiologic saline for injection, 100 ml/bag, q24h, following Ilaprazole Sodium with a time interval of 12 h.
  Arms: Ilaprazole Sodium
Drug: Placebo 2 — Physiologic saline for injection, 100 ml/bag, q12h, dosing on the first day.
  Arms: Esomeprazole Sodium

SUMMARY:
The purpose of this study is to evaluate the efficacy of the study drug (Ilaprazole Sodium for Injection) for potential effect on preventing stress ulcer bleeding in vulnerable population by comparing the radio of upper gastrointestinal bleeding when they are administered Ilaprazole Sodium for Injection and Esomeprazole Sodium for Injection respectively.

ELIGIBILITY:
Inclusion Criteria:

* voluntarily signed informed consent form by subjects per se or their guardians.
* 18-74 years of age, female or male;
* required by the ICU treatment, and is intended to be treated over 72 hours.
* intragastrically intubated for at least 72 hours;
* APACHE II scoring within 15 to 25 (containing upper and lower value)
* intubated by mechanical assistance for breath for intended 48 hours without permission of assistance withdrawal. (Combing clinical observation, patients judged cannot breathing without artificial assistance within 48 hours should meet the any of criteria as following: 1) PEEP > 5; 2) FiO2 > 0.4; 3) Pressure of assisting breathing machine > 13 cmH2O; 4) body temperature over 38℃; 5) CRP ≥ 100 mg/L.
* in addition to mechanical ventilation, at least one major factor that may lead to irritable ulcer bleeding occurred as following within 48 hours prior to random group-assignment.

  1. complex organ surgery at Level 3 or above (surgery duration > 3 hours);
  2. disease history of gastrointestinal ulcer or hemorrhage;
  3. multiple injuries (score (ISS) ≥ 16);
  4. shock
  5. multiple organ dysfunction syndrome (MODS);
  6. sepsis (as per definition of issued by the Society of Critical Care Medicine (SCCM) and European Society of Intensive Care Medicine (ESICM) in 2016)
  7. acidosis (arterial pH < 7.3);
  8. coagulation dysfunction (INR > 1.5, platelets < 50 * 109/L or APTT > 2 times normal value;
  9. coma (GCS ≤ 10);
  10. receiving high dose corticosteroids (over 250 mg/d hydrocortisone or other equivalent dose corticosteroids);
  11. 30%-70% body surface burn;

Exclusion Criteria:

* a history of gastric or esophageal surgery, intestinal obstruction, or hospitalization in the ICU after esophageal, gastric, or duodenal surgery in the past 3 months;
* lesions of the upper digestive tract (e.g., duodenal ulcer, gastric ulcer, acute gastric mucosa lesions, esophageal varices, malignant tumors, etc.) that are known to be likely to bleed, and other evidences indicating gastrointestinal bleeding occurs (esophageal and gastric varices bleeding, duodenal ulcer bleeding);
* hemoglobin < 60g/L (6.0g/dl);
* significant factor indicating bleed occurs during swallowing (such as oral and maxillofacial injuries, hemoptysis, etc.);
* renal failure;
* cardiopulmonary resuscitation conducted during hospitalization period;
* serious liver disease, defined as Child-Pugh C-grade;
* contraindicated for gastric intubation (such as esophageal stenosis);
* pregnancy or pregnancy test showing positive;
* documented or supposed to be hypersensitive to PPIs (Ilaprazole, Esomeprazole, Omeprazole, Lansoprazole, Dextran lansoprazole, Rabeprazole or Pantoprazole);
* participated in other clinical studies within 30 days prior to random assignment;
* use any PPI or treated by H2RA within 12 hours prior to random assignment;
* co-administering or unavoidable using drugs that may interact with Ilaprazole Sodium or Esomeprazole Sodium: e.g., Warfarin (including other vitamin K antagonists), Cisapride, Phenytoin, Atazanavir, Nefenavir, Ritonavir, Saquinavir, Digoxin, Tacrolimus, Methotrexate.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 449 (Actual)
Dates: Start 2021-07-16 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
Preventing clinically significant gastrointestinal bleeding | Day 1 to Day 3
  (1) Bright red blood is observed in gastric tube and not cleared by gavage washing with at least 100mL of standard physiological saline at room temperature for 5 to 10 minutes;
Preventing clinically significant gastrointestinal bleeding | Day 1 and Day 2
  (2) During the Day 1 to Day 2 days of the treatment: If coffee-like substances are observed in the gastric tube, immediately rinse the stomach with at least 100ml of standard physiological saline at room temperature, every 2 hours (± 20 minutes) from the time of first observation, and the coffee-like substances were still observed after 8 hours (the occult blood screening reagent remains positive, and the occult blood result is required to be positive);
Preventing clinically significant gastrointestinal bleeding | Day 3
  (3) On the Day 3 of the treatment - end of treatment: If coffee-like substances are observed in the gastric tube, immediately rinse the stomach with at least 100ml of standard physiological saline at room temperature, once per hour (± 20 minutes), and the coffee-like substances are still observed after 4 hours (occult blood screening reagent continues to be positive, and occult blood results are required to be positive).
Preventing clinically significant gastrointestinal bleeding | Day 1 to Day 3
  (4) Hematemesis or bloody stools originating from the upper gastrointestinal tract (as determined by the researchers, such as tarry stools and positive gastric occult blood).

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shanghai Jiaotong University Affiliate Ruijin Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hopspital of Xinjiang Medical University, Ürümqi, Xinjiang